CLINICAL TRIAL: NCT03164902
Title: Evaluation of Wirelessly Observed Therapy to Optimize Adherence in Patients With Hepatitis C and Increased Risk for Nonadherence to Treatment
Brief Title: Digimeds to Optimize Adherence in Patients With Hepatitis C and Increased Risk for Nonadherence
Acronym: DASH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Proteus Digital Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PB-WOTFORHEPC
Record Dates: First submitted 2017-05-22; First posted 2017-05-24 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Hepatitis C, Chronic; Nonadherence, Patient
MeSH Terms: conditions — Hepatitis C, Chronic; Patient Compliance

STUDY DESIGN:
Masking Description: Sponsor will be blinded from any interim analysis results (except for safety outcomes) until the final analysis. A data monitoring committee has been formed to review interim analyses for study futility and safety.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Digital Medicine Arm (Experimental): Subjects enrolled in this single arm study will be directed to use digital medicine versions of their hepatitis C therapy for the duration of therapy.
  Interventions: Device: Digital Medicine

INTERVENTIONS:
Device: Digital Medicine — The subjects in the study will be monitored using the Proteus Discover offering. Subjects will use Proteus Discover plus a digital version of HCV therapy (IS co-encapsulated with fixed-dose velpatasvir and sofosbuvir; fixed-dose ledipasvir and sofosbuvir; or fixed-dose glecaprevir and pibrentasvir; or fixed-dose sofosbuvir, velpatasvir, and voxilaprevir). The subject's prescribed HCV medication will be co-encapsulated with the Proteus Ingestible Sensor pill by an appropriately licensed and qualified pharmacy as per a licensed health care provider's order (prescription).

SUMMARY:
This study evaluates the ability of digital medicines, Proteus Discover, to promote adherence and thus achieving a cure for hepatitis C in patients at high risk for not adhering to their hepatitis therapy. In this single-arm, prospective study, subjects at high risk for nonadherence will be prescribed hepatitis C therapy that will be co-encapsulated with ingestible sensors (creating the digital medicine) by a pharmacy. Both the subject and the providers will have access to the ingestion adherence.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) is a preventable and curable blood-borne virus. Adherence to HCV therapies is essential to achieve sustained virologic response (SVR) or cure. New direct-acting agents (DAA) are now available, such as fixed-dose combination of ledipasvir and sofosbuvir, which is given once daily with or without ribavirin to treat HCV infection in 8-12 weeks, which can cure hepatitis C with a once daily regimen.

which is given once daily with or without ribavirin to treat HCV infection in 8-12 weeks.

Providers and third-party payers are concerned that patients use these high-cost therapies as prescribed and obtain the intended value of their treatment, so as to prevent otherwise avoidable medicine wastage and re-treatment. Some HCV-infected patients are currently excluded from using the newer direct-acting therapies because they are considered to have a high risk of not completing their intended treatment, or they do not have access to care due to other issues like transportation difficulties.

Additionally, third party payers and providers have proposed to assess patient adherence during treatment with HCV RNA level and additional adherence assessments. However, determining adherence to anti-viral therapy based upon decreases that are observed in RNA titers at intermittent intervals, or periodic assessments of medication use, subsequent to therapy initiation are indirect and retrospective. Additionally, this practice can be a burden for patients, especially those who live far away from their providers.

Proteus Discover™ provides wirelessly observed therapy (WOT) for passive direct, timely confirmation of medication ingestion. Proteus Discover includes a FDA cleared and CE-marked device, which consists of three components: 1) an Ingestible Sensor (IS) embedded inside of a placebo pill, which can be co-encapsulated with prescribed medication (CEM); 2) a wearable sensor patch (herein referred to as the Proteus Patch), which passively detects and stores time-stamped CEM ingestions, as well as physiological and behavioral metrics such as heart rate and activity patterns (e.g., step count, time spent in physical activity, number of hours of rest); and 3) software to aggregate and display Proteus Patch data. The offering also includes the Proteus Discover App, which allows the subject to review and interact with the data via a mobile device. Providers can view the data via the Proteus Discover Portal.

To provide WOT in this study, the Proteus Ingestible Sensor pill will be placed in a capsule along with HCV medication by the patient's pharmacy to create a digital medicine version of the therapy. The adhesive wearable sensor patch worn by the patient on the left lower torso will be used for detection of CEM ingestions which are then displayed on a mobile application for the patient, and on a web portal for physicians and the study healthcare teams to assist them in identifying when support for the subject may be needed for taking medication consistently.

ELIGIBILITY:
Participants must have insurance or other method (e.g. patient assistance program) to pay for medicine.

Inclusion Criteria:

* A subject must meet ALL of the following criteria to be considered for enrollment into this study:

  1. Adults (≥18 years old) who are diagnosed with hepatitis C deemed chronic by the investigator
  2. Candidate for treatment for oral direct acting agent for hepatitis C such as fixed-dose velpatasvir and sofosbuvir; fixed-dose ledipasvir and sofosbuvir; or fixed-dose glecaprevir and pibrentasvir with insurance coverage for therapy. Subjects may take other medicines that will not be co-encapsulated (e.g. ribavirin)
  3. One of more of the following risk factors for nonadherence:

     1. Active alcohol or substance abuse (positive urine drug screen, illicit use in past 3 months, and/or in opioid substitution program), OR
     2. Patient reported history of hospitalization within past 2 years for a psychiatric comorbidity, OR
     3. Evidence of nonadherence to medications (e.g. self-report or refill history indicative of nonadherence), OR
     4. History of at least one missed clinic visit for hepatitis management, OR
     5. Patient-reported history of one or more transportation barriers (e.g. burden due to time and/or distance or lack of access to regular transportation) to healthcare access, which creates a risk for missed or delayed care
  4. Study subject has daily access to a telephone for communicating with the study personnel and study personnel contacting the study subject
  5. Ability to read and understand the instructions for the study.
  6. Willingness to adhere to all study procedures (both onsite and offsite), including troubleshooting of the product by a third-party, if needed.
  7. Capacity to and willing to provide informed consent. All subjects must have a signed informed consent document prior to participating in this study
  8. Currently owns and uses a smart phone or tablet, or has capacity to learn use of study mobile device as determined by investigator.
  9. Adequate data connectivity at home via cellular service and/or access to a secure wireless internet (WiFi) network with the proficiency to connect a mobile device to the WiFi network.

     * Note: None of the five individual sub-criteria (i.e., 3a, 3b, 3c, 3d, or 3e) alone may be used to qualify more than approximately 20% of the total study population for randomization. For example, "3d" may be used to qualify no more than 20% of the study population for randomization without an additional sub-criteria also being met (e.g., "3d" + "3a"). The data center will monitor the use of these five enrolment sub-criteria, and study sites will be notified when qualification for enrollment may no longer be based upon meeting only a specific one of the five sub-criteria alone (e.g., "3d" alone).

Exclusion Criteria:

* ANY 1 of the following will exclude a subject from being enrolled into the study:

  1. BMI > 40 kg/m2 2. Active skin infection or active dermatitis, OR history of chronic inflammatory skin condition including psoriasis and chronic dermatitis (except atopic dermatitis) 3. Allergy to adhesive bandages/tapes (e.g. Band-Aids®) 4. Severely decompensated cirrhosis (Child-Pugh C) or a liver transplant candidate 5. Any condition that in the investigator's opinion could preclude safe participation in the study (e.g. contraindication to hepatitis C therapy) or would preclude the subject from being able to participate in the study protocol requirements 6. Participating in a drug study or medical device clinical study (including its safety follow-up period as defined by protocol) 30 days prior to study start or completion 7. Unwilling to take a gelatin capsule because it is manufactured from animal origins (e.g. for religious reasons) 8. Allergy to food dye 10. Terminal illness (≤ 1 year of life anticipated). 10. Currently known to be pregnant or nursing an infant. 11. For women of childbearing potential, not using an acceptable form of contraception for at least 2 months prior to screening and throughout the duration of the study. Accepted means of contraception include oral contraceptive or implant, condom, diaphragm, spermicide, intrauterine device, tubal ligation, or partner with vasectomy.

  12. Positive pregnancy test during screening 13. Inability to swallow the test capsule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Estimated)
Dates: Start 2017-07-21 (Actual); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
SVR12 Rate | 12 weeks following completion of their hepatitis C therapy
  Proportion of subjects achieving sustained viral response, 12 weeks following completion of their hepatitis C therapy

SECONDARY OUTCOMES:
SVR4 Rate | 4 weeks following completion of their hepatitis C therapy
  Proportion of subjects achieving sustained viral response, 4 weeks following completion of their hepatitis C therapy
Ingestion Adherence | 8 to 16 weeks (during therapy)
  Mean ingestion adherence to the primary hepatitis C therapy measured by the digital medicine offering
Safety Profile:Summary details of all adverse events during the study | Up to 24 weeks
  Summary details of all adverse events during the study
Subject Satisfaction | 4 weeks following completion of their hepatitis C therapy
  Feedback from subjects during the study via a survey form

OTHER OUTCOMES:
Treatment efficiency | Up to 24 weeks
  Number of clinic and lab visits and other resources used during the study

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sulkowski, MD, Principal Investigator — Johns Hopkins University
Locations (16):
- United States (16):
  - University of Alabama, Birmingham, Alabama
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Denver Health, Denver, Colorado
  - Providence Health System, Washington D.C., District of Columbia
  - Orlando Immunology Center, Orlando, Florida
  - Apex Clinical Research, Tampa, Florida
  - The Ruth M. Rothstein CORE Center, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - The Research Institute, Springfield, Massachusetts
  - Harper University Hospital, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Southwest Care Center, Santa Fe, New Mexico
  - Duke University Medical Center, Durham, North Carolina
  - Harborview Medical Center, Seattle, Washington
  - SSM Health Dean Medical Group, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Armstrong GL, Wasley A, Simard EP, McQuillan GM, Kuhnert WL, Alter MJ. The prevalence of hepatitis C virus infection in the United States, 1999 through 2002. Ann Intern Med. 2006 May 16;144(10):705-14. doi: 10.7326/0003-4819-144-10-200605160-00004. PMID 16702586
- [Background] Younossi ZM, Park H, Gordon SC, Ferguson JR, Ahmed A, Dieterich D, Saab S. Real-world outcomes of ledipasvir/sofosbuvir in treatment-naive patients with hepatitis C. Am J Manag Care. 2016 May;22(6 Spec No.):SP205-11. PMID 27266950
- [Derived] Sulkowski M, Luetkemeyer AF, Wyles DL, Martorell C, Muir A, Weisberg I, Gordon SC, McLain R, Huhn G. Impact of a digital medicine programme on hepatitis C treatment adherence and efficacy in adults at high risk for non-adherence. Aliment Pharmacol Ther. 2020 Jun;51(12):1384-1396. doi: 10.1111/apt.15707. Epub 2020 Apr 30. PMID 32352586